CLINICAL TRIAL: NCT04925206
Title: A Multicenter, Open Label Phase 1 Study to Evaluate the Safety and Efficacy of a Single Dose of Autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (hHSPCs) in Subjects with Transfusion Dependent Β-Thalassaemia
Brief Title: A Safety and Efficacy Study Evaluating ET-01 in Subjects with Transfusion Dependent Β-Thalassaemia
Acronym: ET-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development plan change
Sponsor: EdiGene (GuangZhou) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-001
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Transfusion Dependent Beta-Thalassaemia
Keywords: Beta-Thalassaemia; CRISPR-Cas9; Human Hematopoietic Stem and Progenitor Cells
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ET-01 (Experimental)
  Interventions: Biological: ET-01

INTERVENTIONS:
Biological: ET-01 — Recruited participants will receive ET-01 IV infusion following myeloablative conditioning with busulfan.

SUMMARY:
This is a single-arm, open label, multi-center, single-dose phase 1 study in subjects with transfusion dependent β-thalassaemia. The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (hHSPCs) using ET-01.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects and/or legal representative fully understand and voluntarily sign informed consent forms.
* Diagnosis of transfusion dependent β-thalassemia (β-TDT) as defined by protocol.
* Be not appropriate to receive conventional allogeneic hematopoietic stem cell transplantation.
* Lansky/Karnofsky score ≥ 70%.
* Eligible for hematopoietic stem cell transplantation and conditioning with busulfan as per investigator's judgement.

Other protocol defined inclusion criteria may apply.

Key Exclusion Criteria:

* Subjects with associated α-thalassemia.
* Subjects with any clinically significant acute or uncontrolled infections.
* History of uncontrolled epilepsy or other mental disorders.
* Previous treatment with allogeneic bone marrow transplantation or gene therapy.

Other protocol defined exclusion criteria may apply.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of collected AEs & SAEs | Within 24 months after ET-01 infusion
All-cause mortality | From signing of informed consent up to 24 months post-ET-01 infusion
Incidence of transplant-related mortality | From baseline (pre-transfusion) up to 12 months post-ET-01 infusion
Total lymphocyte count | Within 24 months after ET-01 infusion
Proportion of subjects with abnormal proliferation of blood cells | Within 24 months after ET-01 infusion

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No